CLINICAL TRIAL: NCT02326909
Title: a Prospective In-vivo Human Study to Assess the Diagnostic Accuracy of Optical Coherence Tomography for Diagnosis and Staging of Upper Urinary Tract Urothelial Carcinoma
Brief Title: Diagnostic Accuracy of Optical Coherence Tomography in Upper Urinary Tract Urothelial Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, M.T.J. Bus, M.D., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL42100.018.12
Record Dates: First submitted 2014-02-05; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Transitional Cell Carcinoma of Urinary Tract
Keywords: Upper Urinary Tract; Optical Coherence Tomography; Transitional Cell Carcinoma; Urothelial Cell Carcinoma; Diagnostic accuracy
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- optical coherence tomography (Experimental): A single 1300 nm OCT measurement will be performed during ureterorenoscopy in patients with upper urinary tract tumour(s)
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Optical Coherence Tomography — Single Optical Coherence Tomography measurement of upper urinary tract tumour taken during ureterorenoscopy
Device: Optical Coherence Tomography — A single 1300 nm OCT measurement will be performed during ureterorenoscopy in patients with upper urinary tract tumour(s)
  Other Names: 1300 nm Optical Coherence Tomography

SUMMARY:
The purpose of this study is to establish in vivo sensitivity and specificity of OCT in the diagnosis of Upper Urinary Tract Urothelial Carcinoma.

DETAILED DESCRIPTION:
Minimal invasive endoscopic treatment for Upper Urinary Tract Urothelial Carcinoma (UUT-UC) has been accepted as a treatment option instead of radical nephroureterectomy for patients with low grade, low stage disease. For this reason, information on tumour stage and grade is important for a clinical decision. Until now,diagnostic ureterorenoscopy combined with histology/cytology is the gold standard. Unfortunately, histology/cytology is often inconclusive.

Optical Coherence Tomography is a new high resolution imaging technique that has potential to provide the urologist real time per-operative information of grade and stage of the disease.

In this study the investigators aim to establish in vivo sensitivity and specificity of OCT in the diagnosis of Upper Urinary Tract Urothelial Carcinoma. Secondary objectives are inter-observer variability of 1300 nm OCT in the diagnosis of UUT-UC and optical properties of cancerous and healthy ureter and collecting system tissue in vivo in humans.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for diagnostic or therapeutic ureterorenoscopy
* Signed informed consent

Exclusion Criteria:

* No signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity of 1300nm OCT in grading and staging UUT-UC | up to 10 minutes
  Only a single OCT measurement will be done during surgery. This measurement will take a maximum of 10 minutes, including preparation of the OCT device
Specificity of 1300nm OCT in grading and staging UUT-UC | up to 10 minutes
  Only a single OCT measurement will be done during surgery. This measurement will take a maximum of 10 minutes, including preparation of the OCT device

OTHER OUTCOMES:
Optical properties of cancerous and healthy ureter and collecting system tissue | up to 10 minutes
  only a single OCT measurement will be done during surgery. This measurement will take a maximum of 10 minutes, including preparation of the OCT device

CONTACTS AND LOCATIONS:
Overall Officials: Jean J. de la Rosette, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Result] Bus MT, Muller BG, de Bruin DM, Faber DJ, Kamphuis GM, van Leeuwen TG, de Reijke TM, de la Rosette JJ. Volumetric in vivo visualization of upper urinary tract tumors using optical coherence tomography: a pilot study. J Urol. 2013 Dec;190(6):2236-42. doi: 10.1016/j.juro.2013.08.006. Epub 2013 Aug 13. PMID 23954585